CLINICAL TRIAL: NCT05940610
Title: The Safety and Efficacy of Mesenchymal Stem Cells-Derived Extracellular Vesicles (MSC-EV) in Acute/Acute-on-Chronic Liver Failure：a Prospective, Randomized, Controlled Clinical Study
Brief Title: The Safety and Efficacy of MSC-EVs in Acute/Acute-on-Chronic Liver Failure
Status: Withdrawn | Phase: Phase 1 / Phase 2 | Type: Interventional
Why Stopped: The supply of msc-ev has been delayed and approval by the Ethics committee will take some time.
Sponsor: Third Affiliated Hospital, Sun Yat-Sen University (Other)
Responsible Party: Principal Investigator, Yang Yang, Head of Department of Hepatic Surgery and Liver Transplantation Center of the Third Affiliated Hospital, Organ Transplantation Institute, Sun Yat-sen University, Third Affiliated Hospital, Sun Yat-Sen University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: MSC-EVs-2 of ThirdSunYatSen
Record Dates: First submitted 2023-07-02; First posted 2023-07-11 (Actual); Last update posted 2023-10-12 (Actual); Status verified 2023-10

CONDITIONS: Acute-On-Chronic Liver Failure; Acute Liver Failure
Keywords: MSC-EVs; Acute-on-chronic liver failure; Acute liver failure; Liver transplantation
MeSH Terms: conditions — Acute-On-Chronic Liver Failure; Liver Failure, Acute

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- MSC-EV group (Experimental): On the basis of standard medical treatment, an additional injection of MSC-EVs will be received by participants once a week for 4 weeks while hospitalized.
  Interventions: Biological: MSC-EVs
- Non-MSC-EV group (No Intervention): In the non-MSC-EV group, patients will receive standard medical treatment and 100ml saline as a control.

INTERVENTIONS:
Biological: MSC-EVs — 10 E10 MSC-EV particles per 100ml for a single dose. Once a week for 4 weeks.
  Arms: MSC-EV group

SUMMARY:
Acute-on-chronic liver failure (ACLF) refers to a liver failure syndrome in which some patients with chronic liver disease with relatively stable liver function suffer from acute liver decompensation and liver failure due to the effects of various acute injury factors，while acute liver failure (ALF) refers to a potentially reversible disorder that was the result of severe liver injury, with an onset of encephalopathy within 8 weeks of symptom appearance and in the absence of pre-existing liver disease. Liver transplantation is the only curative treatment for this type of end-stage liver disease, but the rapid disease progression and lack of donors limit its application. The potential of MSCs to repair or regenerate damaged tissue and suppress immune responses makes them promising in the treatment of liver diseases, especially in the field of liver transplantation. Many studies have shown that MSC-based therapies can reduce the symptoms of liver disease due to their paracrine effects. It has been confirmed in previous studies that infusion of allogeneic MSCs is safe and convenient for patients with ACLF and improve liver function and decrease the incidence of severe infections. Compared to the cells they derive from, mesenchymal stem cells-derived extracellular vesicles (MSC-EVs) are gradually gaining attention for their enhanced safety, as they do not replicate or cause microvascular embolism, and can be easily stored without losing their properties. It represents a novel and effective cell-free therapeutic agent as alternative to cell-based therapies for liver diseases, and liver failure was also concerned. This study was designed to evaluate the safety and efficacy of MSC-EVs in ACLF/ALF .

DETAILED DESCRIPTION:
In the MSC-EV group (experimental group), onthe basis of standard medical treatment, 10 patients will receive a single injection of MSC-EV . In the non-MSC-EV group (control group), 10 patients will not receive MSC-EV therapy but standard medical treatment. The standard medical treatment iclude nutritional supplementation, administration of human serum albumin and fresh frozen plasma, anti-viral therapy (if hepatitis virus-related ACLF/ALF), liver protective treatment and other appropriate treatment for complications.

The outcome of the experimental group will be compared with that of similar control patients who will not receive MSC-EV. Both of the two groups will receive standard medical treatment. Patients participated in the experimental cohort will be infused with a single dose of 10 E10 MSC-EV particles per 100ml, when they are inpatient.

ELIGIBILITY:
Inclusion Criteria:

* aged 18-65 years old;
* Acute on chronic liver failure-which is characterized by acute hepatic insult manifesting as jaundice (serum total bilirubin [TBil] ≥ 10×ULN umol/L) and coagulopathy (international normalized ratio [INR] ≥ 1.5 or prothrombin activity < 40%), complicated within 4 weeks by ascites and/or encephalopathy as determined by physical examination, in patients with previously diagnosed or undiagnosed chronic liver disease; Acute liver failure-a potentially reversible disorder that was the result of severe liver injury, with an onset of encephalopathy within 8 weeks of symptom appearance and in the absence of pre-existing liver disease.
* Total bilirubin (TBil) ≥ 171umolL or daily increase ≥17.1umol/L;
* Prothrombin activity (PTA) between 20% and 40% (or INR between 1.5 and 2.6);
* No hepatic encephalopathy, or encephalopathy below grade II (including grade II);

Exclusion Criteria:

* Patients with primary or metastatic liver cancer
* Severe active bleeding or diffuse intravascular coagulation
* Patients who are allergic to blood products or drugs used in treatment, such as plasma, heparin and protamine;
* MELD score >30
* Other serious disease including heart disease, lung disease, blood disease, autoimmune disease, diabetes, active uncontrolled infection,etc.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2023-09-01 (Estimated); Primary Completion 2024-09-30 (Estimated); Study Completion 2025-10-01 (Estimated)

PRIMARY OUTCOMES:
Number of participants with MSC-EV infusion-related toxicity as assessed by CTCAE v4.0. | 24 hours after injection
  Incidence, timing and severity of any clinical complication related to MSC-EV infusion, such as tympanic body temperature, heart rate, mean arterial blood pressure and allergy, as assessed by CTCAE v4.0 .
Aspartate aminotransferase (AST) | 6 months after first rejection
  Collect clinical results reflecting liver function
Alanine aminotransferase (ALT) | 6 months after first rejection
  Collect clinical results reflecting liver function
Bilirubin level | 6 months after first rejection
  Collect clinical results reflecting liver function
International normalized ratio (INR) | 6 months after first rejection
  Collect clinical results reflecting liver function
Carbohydrate Compound antigen (GGT) level | 6 months after first rejection
  Collect clinical results reflecting liver function
Adverse events | 6 months after first rejection
  Any adverse events which may related to MSC-EV infusion

SECONDARY OUTCOMES:
Number of survived patients at 1 year, according to the follow-up results | 12 months
  Patients who are surviving, as assessed by outpatient or telephone follow-up, at 1 year after rejection
Proportion of immune cell subsets from biopsy or blood samples ,at months 1-6 after infusion. | 6 months
  A series of immune cell subsets will be analyzed, including T cells (CD3+), CD4+ T cells (CD3+ CD4+ lymphocytes), CD8+ T cells (CD3+ CD8+ lymphocytes), naïve CD4+ T cells (CD4+ CD45RAhigh lymphocytes), memory CD4+ T cells (CD4+ CD45RO+ lymphocytes), natural killer (NK) cells (CD3- CD56+ lymphocytes), as well as B cells (CD19+ lymphocytes)

CONTACTS AND LOCATIONS:
Locations (1):
- Third Affiliated Hospital, Sun Yat-Sen University, Guangzhou, Guangdong, China